CLINICAL TRIAL: NCT00001013
Title: A Randomized, Comparative, Double-Blind Trial of Trimetrexate (CI-898) With Leucovorin Calcium Rescue Versus Trimethoprim / Sulfamethoxazole for Moderately Severe Pneumocystis Carinii Pneumonia in Patients With AIDS
Brief Title: Comparison of Trimetrexate Plus Leucovorin Calcium Rescue Versus Sulfamethoxazole-Trimethoprim in the Treatment of Pneumocystis Carinii Pneumonia (PCP) in Patients With AIDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 029; 11005 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimethoprim-Sulfamethoxazole Combination; Trimetrexate; AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Pentamidine; Infusions, Intravenous; Leucovorin; Drug Therapy, Combination; Folic Acid Antagonists; Aerosols; Acquired Immunodeficiency Syndrome; Antiprotozoal Agents; AIDS-Related Complex; Sulfamethoxazole-Trimethoprim
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — trimetrexate glucuronate; Pentamidine; Trimethoprim, Sulfamethoxazole Drug Combination; Leucovorin

INTERVENTIONS:
Drug: Trimetrexate glucuronate
Drug: Pentamidine isethionate
Drug: Sulfamethoxazole-Trimethoprim
Drug: Leucovorin calcium

SUMMARY:
To compare the safety and effectiveness of an investigational drug therapy (trimetrexate plus leucovorin calcium) with that of conventional therapy (sulfamethoxazole-trimethoprim) in the treatment of moderately severe Pneumocystis carinii pneumonia (PCP) in patients who have AIDS, are HIV positive, or are at high risk for HIV infection.

DETAILED DESCRIPTION:
New treatments are needed to reduce the mortality rate from PCP in AIDS patients and to reduce the high relapse rate found after conventional therapy. Trimetrexate (TMTX) was chosen for this trial because it was found to be much more potent than sulfamethoxazole/trimethoprim (SMX/TMP) against the PCP organism in laboratory tests. Also TMTX, in combination with leucovorin (LCV), did not cause severe toxicity in a preliminary trial. It is believed that TMTX will be more effective than SMX/TMP in treating PCP and in preventing a recurrence of PCP. Preliminary studies suggest that aerosolized pentamidine (PEN) is likely to be effective in preventing a recurrence of PCP.

Patients entered in the study are randomly assigned to TMTX / LCV or to SMX/TMP for a 21-day trial. For the first 10 days, the trial is double-blind (neither patient nor physician knows which drugs the patient is receiving), and drugs are given by intravenous infusion. TMTX is given once every 24 hours and LCV every 6 hours; SMX/TMP is given every 6 hours. Doses are determined by body size. After the first 10 days, LCV and SMX/TMP may be given orally. Doses are adjusted or treatment is changed to intravenous PEN if side effects are too severe. During the 21-day trial, zidovudine (AZT) may not be used because of possible increased bone marrow toxicity. AZT may be resumed as soon as the patient's white cell count is acceptable. Aerosolized PEN therapy is begun 7 - 10 days after completion of therapy for the acute episode. PEN is inhaled once weekly for 4 weeks, then every 2 weeks for 48 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Acetaminophen:
* 650 mg prescribed as necessary for temperature > 38.7 degrees C. Acetaminophen should not be prescribed as a standing order for more than 48 hours.

Prior Medication:

Allowed:

* Zidovudine (AZT) as long as such therapy is suspended prior to randomization and not reinstituted until therapy for the acute episode is completed and the patient's white blood cell count is acceptable.
* Other myelosuppressive therapies which may be handled in the same manner as AZT.
* Prophylaxis for Pneumocystis carinii pneumonia (PCP).
* Unequivocal diagnosis of Pneumocystis carinii pneumonia (PCP) by morphologic confirmation of three or more typical P. carinii organisms in sputum, bronchoalveolar lavage fluid, or lung tissue obtained by transbronchial or open-lung biopsy within 3 days before or after randomization. If morphologic confirmation is not possible prior to therapy, patients may be randomized if the investigator believes there is a high suspicion of PCP based on clinical presentation. If morphologic diagnosis cannot be established within 6 days of randomization, the patient will be withdrawn from study therapy. Resting (A-a) DO2 < 30 torr on room air. Patient, parent, guardian, or person with power of attorney gives informed consent.

Exclusion Criteria

Co-existing Condition:

Patients will be excluded for the following reasons:

* History of Type I hypersensitivity (i.e., urticaria, angioedema, or anaphylaxis), exfoliative dermatitis, or other life-threatening reaction secondary to antibiotics containing sulfa, trimethoprim, or trimetrexate.
* History of life-threatening pentamidine toxicity.

Concurrent Medication:

Excluded:

* Other drugs for the treatment or prevention of AIDS or Pneumocystis carinii pneumonia (PCP).
* Disalcid.
* Aspirin.
* Acetaminophen q4h as a standing order for more than 48 hours.

Prior Medication:

Excluded within 14 days of study entry:

* Systemic steroids exceeding physiological replacement.
* Other investigational drugs including ganciclovir.
* Excluded within 6 weeks of study entry:
* Another antiprotozoal regimen for this episode for therapy of active Pneumocystis carinii pneumonia (PCP).
* Patients who are unable to have arterial blood gas analysis (ABG's) on room air.
* Patients for whom a liter of intravenous fluid (5 percent dextrose in water) per 24 hours, which is required to maintain blinding, would be medically inadvisable.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 364
Dates: Study Completion 1991-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sattler FR, Study Chair
Locations (23):
- United States (23):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Northwestern Univ Med School, Chicago, Illinois
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Louisiana State Univ Med Ctr / Tulane Med School, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Univ of Massachusetts Med Ctr, Worcester, Massachusetts
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - City Hosp Ctr at Elmhurst / Mount Sinai Hosp, Elmhurst, New York
  - Beth Israel Med Ctr / Peter Krueger Clinic, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - SUNY - Stony Brook, Stony Brook, New York
  - SUNY / State Univ of New York, Syracuse, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Holmes Hosp / Univ of Cincinnati Med Ctr, Cincinnati, Ohio
  - Univ Hosp of Cleveland / Case Western Reserve Univ, Cleveland, Ohio
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Thomas Jefferson Med College, Philadelphia, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina

REFERENCES:
- [Background] Sattler FR, Frame P, Davis R, Nichols L, Shelton B, Akil B, Baughman R, Hughlett C, Weiss W, Boylen CT, et al. Trimetrexate with leucovorin versus trimethoprim-sulfamethoxazole for moderate to severe episodes of Pneumocystis carinii pneumonia in patients with AIDS: a prospective, controlled multicenter investigation of the AIDS Clinical Trials Group Protocol 029/031. J Infect Dis. 1994 Jul;170(1):165-72. doi: 10.1093/infdis/170.1.165. PMID 8014493